CLINICAL TRIAL: NCT04971148
Title: Correlation of Peak Tidal Inspiratory Flow Measured Before and After Extubation in Adult Patients With Hypoxemia, and Patients' Responses to Different Flows Above Their Peak Tidal Inspiratory Flow During High Flow Nasal Cannula Therapy
Brief Title: Correlation of Peak Tidal Inspiratory Flow Measured Before and After Extubation in Adult Patients With Hypoxemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: Rush University Medical Center (Other)
Collaborators: Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HFNC-Flow-004
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hypoxemic Respiratory Failure
Keywords: high-flow nasal cannula; flow setting; peak tidal inspiratory flow; hypoxemia
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive different HFNC flow settings (matching their peak tidal inspiratory flow [PTIF], 1.33 times of PTIF, 1.67 times of PTIF and 2 times of PTIF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HFNC flow set at patient peak tidal inspiratory flow (Active Comparator): HFNC flow will be set at the level that matches patient peak tidal inspiratory flow
  Interventions: Other: HFNC flow set at patient peak tidal inspiratory flow
- HFNC flow set at 1.33 times of patient peak tidal inspiratory flow (Experimental): HFNC flow will be set at the level that is 1.33 times of patient peak tidal inspiratory flow
  Interventions: Other: HFNC flow set at 1.33 times of patient peak tidal inspiratory flow
- HFNC flow set at 1.67 times of patient peak tidal inspiratory flow (Experimental): HFNC flow will be set at the level that is 1.67 times of patient peak tidal inspiratory flow
  Interventions: Other: HFNC flow set at 1.67 times of patient peak tidal inspiratory flow
- HFNC flow set at 2 times of patient peak tidal inspiratory flow (Experimental): HFNC flow will be set at the level that is 2 times of patient peak tidal inspiratory flow
  Interventions: Other: HFNC flow set at 2 times of patient peak tidal inspiratory flow

INTERVENTIONS:
Other: HFNC flow set at patient peak tidal inspiratory flow — HFNC flow will be set at the level equal to patient peak tidal inspiratory flow
  Arms: HFNC flow set at patient peak tidal inspiratory flow
Other: HFNC flow set at 1.33 times of patient peak tidal inspiratory flow — HFNC flow will be set at 1.33 times of patient peak tidal inspiratory flow
  Arms: HFNC flow set at 1.33 times of patient peak tidal inspiratory flow
Other: HFNC flow set at 1.67 times of patient peak tidal inspiratory flow — HFNC flow will be set at 1.67 times of patient peak tidal inspiratory flow
  Arms: HFNC flow set at 1.67 times of patient peak tidal inspiratory flow
Other: HFNC flow set at 2 times of patient peak tidal inspiratory flow — HFNC flow will be set 2 times of patient peak tidal inspiratory flow
  Arms: HFNC flow set at 2 times of patient peak tidal inspiratory flow

SUMMARY:
In this study, patients who are ready for extubation and indicated for high-flow nasal cannula therapy after extubation will be enrolled, the investigators would measure the patient peak tidal inspiratory flow (PTIF) pre and post extubation to explore the correlation between the two PTIFs. Moreover, different HFNC flows would be applied, to explore the patient response in terms of oxygenation and lung aeration to different flow ratios that matched and are above post-extubation PTIF.

DETAILED DESCRIPTION:
High-flow nasal cannula (HFNC) oxygen therapy has been shown to improve oxygenation, reduce the need for intubation for patients with acute hypoxemic respiratory failure (AHRF) and avoid reintubation for post-extubation patients who had high-risk factors. HFNC refers to the delivery of gas at flows that exceed the patient peak inspiratory flow during tidal breathing, However, patient peak tidal inspiratory flow (PTIF) is found to vary greatly among different patients, from 20 to 50 L/min, making it difficult to properly set HFNC in a way to achieve the desired effects. In two recently published studies in intubated patients, PTIF varied from 25-65 L/min or 40-80 L/min, thus this study aims to investigate the correlation between pre-extubation PTIF in different modalities of SBT and post-extubation PTIF for adult patients, who are indicated to use HFNC immediately after extubation. In addition, the investigators aim to explore the patient response in terms of oxygenation and lung aeration to different flow ratios that matched and are above post-extubation PTIF.

ELIGIBILITY:
Inclusion Criteria:

* Adult intubated patients aged between 18 to 90 years
* Pass spontaneous breathing trial and receive the order to be extubated
* Have at least one of the indications to use HFNC after extubation

Exclusion Criteria:

* Need to use inhaled epoprostenol via HFNC
* Pregnant
* Unable to use resuscitation mask, such as facial trauma, claustrophobia
* Non-English speaker
* Inability to verbally communicate
* Using extracorporeal membrane oxygenation (ECMO)
* Hemodynamically unstable
* Difficult airway

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
SpO2/FIO2 | 20 minutes after each flow setting
  Twenty mins after each flow setting, pulse oximetry divided by fraction of inspired oxygen will be used to assess patient's oxygenation response to different flow

SECONDARY OUTCOMES:
End-expiratory lung volume assessed by EIT | 20 minutes after each flow setting
  Twenty mins after each flow setting, electrical impedance tomography (EIT) will be used to assess patient's end -expiratory lung volume 20 mins after each flow setting
self-evaluated comfort | 20 minutes after each flow setting
  Twenty mins after each flow setting, patient comfort will be assessed using a visual numerical scale with a score of 0 as the worst and 10 as the best comfort

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, PhD, Principal Investigator — Rush University
Locations (2):
- Rush university medical center, Chicago, Illinois, United States
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data will be shared upon reasonable request 3 months after publication.
Supporting Information: Study Protocol, ICF
Time Frame: 3 months after the study is published
Access Criteria: the investigators need to send their IRB approved research protocol to Jie_li@rush.edu

REFERENCES:
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Rochwerg B, Granton D, Wang DX, Helviz Y, Einav S, Frat JP, Mekontso-Dessap A, Schreiber A, Azoulay E, Mercat A, Demoule A, Lemiale V, Pesenti A, Riviello ED, Mauri T, Mancebo J, Brochard L, Burns K. High flow nasal cannula compared with conventional oxygen therapy for acute hypoxemic respiratory failure: a systematic review and meta-analysis. Intensive Care Med. 2019 May;45(5):563-572. doi: 10.1007/s00134-019-05590-5. Epub 2019 Mar 19. PMID 30888444
- [Background] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464
- [Background] Hernandez G, Vaquero C, Gonzalez P, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Colinas L, Cuena R, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Conventional Oxygen Therapy on Reintubation in Low-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Apr 5;315(13):1354-61. doi: 10.1001/jama.2016.2711. PMID 26975498
- [Background] Yasuda H, Okano H, Mayumi T, Narita C, Onodera Y, Nakane M, Shime N. Post-extubation oxygenation strategies in acute respiratory failure: a systematic review and network meta-analysis. Crit Care. 2021 Apr 9;25(1):135. doi: 10.1186/s13054-021-03550-4. PMID 33836812
- [Background] Butt S, Pistidda L, Floris L, Liperi C, Vasques F, Glover G, Barrett NA, Sanderson B, Grasso S, Shankar-Hari M, Camporotaa L. Initial setting of high-flow nasal oxygen post extubation based on mean inspiratory flow during a spontaneous breathing trial. J Crit Care. 2021 Jun;63:40-44. doi: 10.1016/j.jcrc.2020.12.022. Epub 2020 Dec 27. PMID 33621890
- [Background] Mauri T, Spinelli E, Dalla Corte F, Scotti E, Turrini C, Lazzeri M, Alban L, Albanese M, Tortolani D, Wang YM, Spadaro S, Zhou JX, Pesenti A, Grasselli G. Noninvasive assessment of airflows by electrical impedance tomography in intubated hypoxemic patients: an exploratory study. Ann Intensive Care. 2019 Jul 22;9(1):83. doi: 10.1186/s13613-019-0560-5. PMID 31332551
- [Background] Mauri T, Alban L, Turrini C, Cambiaghi B, Carlesso E, Taccone P, Bottino N, Lissoni A, Spadaro S, Volta CA, Gattinoni L, Pesenti A, Grasselli G. Optimum support by high-flow nasal cannula in acute hypoxemic respiratory failure: effects of increasing flow rates. Intensive Care Med. 2017 Oct;43(10):1453-1463. doi: 10.1007/s00134-017-4890-1. Epub 2017 Jul 31. PMID 28762180
- [Result] Li J, Jing G, Scott JB. Year in Review 2019: High-Flow Nasal Cannula Oxygen Therapy for Adult Subjects. Respir Care. 2020 Apr;65(4):545-557. doi: 10.4187/respcare.07663. PMID 32213602
- [Result] Li J, Scott JB, Fink JB, Reed B, Roca O, Dhand R. Optimizing high-flow nasal cannula flow settings in adult hypoxemic patients based on peak inspiratory flow during tidal breathing. Ann Intensive Care. 2021 Nov 27;11(1):164. doi: 10.1186/s13613-021-00949-8. PMID 34837553